CLINICAL TRIAL: NCT02824133
Title: A Phase I/II, Open-Label, Multicentre Study to Assess The Safety, Tolerability, Pharmacokinetics and Clinical Efficacy of AZD4547 in Patients With Relapsed/Refractory Glioma Positive for an FGFR Fusion
Brief Title: Treatment With AZD4547 for Recurrent Malignant Glioma Expressing FGFR-TACC Gene Fusion"
Acronym: TARGET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140402; 2014-005428-81 (EudraCT Number)
Record Dates: First submitted 2015-12-21; First posted 2016-07-06 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-04

CONDITIONS: Recurrent IDHwt Gliomas With FGFR3-TACC3 Fusion; Recurrent IDHwt Gliomas With FGFR1-TACC1 Fusion
Keywords: Glioma grade III; Glioma grade IV; Glioma recurrent; IDHwt; FGFR-TACC fusion
MeSH Terms: interventions — AZD4547; Enzymes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD4547 (Experimental): AZD4547: intake of 80mg bd (160mg/day), on a continuous schedule.
  Interventions: Drug: AZD4547

INTERVENTIONS:
Drug: AZD4547 — 80 mg bd (per os)
  Other Names: Potent and selective inhibitor of FGFR-1, 2 and 3 receptor tyrosine kinases (enzyme and cellular phosphorylation endpoints) with lower potency for inhibition of IGF1R and KDR

SUMMARY:
The investigators will look for the presence of the fusion gene in all patients operated on for glioma. This search will be limited to all gliomas that show no IDH1 mutation, the latter being sought in both routine and anomalies never co-existing.

The hypothesis is that the rate of progression-free survival in grade IV gliomas and III without IDH1 mutation, with the usual chemotherapy, only 15% at 6 months (ie, 85% of patients relapse before 6 months of treatment), must be with this new treatment 35% (primary endpoint).

The main objective is the evaluation of disease-free survival at 6 months.

DETAILED DESCRIPTION:
3% of GBM and IDHwt gliomas have a highly oncogenic FGFR-TACC gene fusion that confers high sensitivity to FGFR inhibitors to tumor cells, in vitro and in vivo. Preclinical data shows that expression of FGFR-TACC fusions confers sensitivity to FGFR inhibitors (including AZD4547) to GBM models.AZD4547 (AstraZeneca) is a potent and selective inhibitor of FGFR-1, 2 and 3 receptor tyrosine kinases. Preclinical data have shown some CNS penetration. Some of the important adverse events are hyperphosphatemia, and ocular complications. The primary objective and assessment criterion is to assess the efficacy of AZD4547 by measuring the rate of Progression Free Survival at 6 months (PFS6) in recurrent malignant glioma patients with FGFR-TACC fusion.Secondary objectives and assessment criteria are: - To characterize the safety, tolerability and PK of AZD4547 in glioma patients

* To further assess the anti-tumor activity of AZD4547 for patients with recurrent glioma with FGFR-TACC fusion based on Overall Response Rate for patients with a measurable residue.
* To further assess the anti-tumor activity of AZD4547 for patients with recurrent glioma with FGFR-TACC fusion based on the duration of PFS
* To further assess the anti-tumor activity of AZD4547 for patients with recurrent glioma with a FGFR-TACC fusion based on Overall Survival AZD4547 Exploratory objectives - To elucidate the mechanism of response and resistance (primary and secondary) by exploratory biomarker analysis Experimental design: This is a phase II study in patients diagnosed with a FGFR3-TACC3 or FGFR1-TACC1 fusion positive glioma presenting with a recurrence of the disease after chemotherapy and radiotherapy. RNA will be systematically screened for the presence of FGFR-TACC in each of the 11 participating centers, and IHC for FGFR3 hyperexpression. The investigators also encourage a wide use of FGFR3 IHC in non participating centers in order to identify additional potential candidates who can be referred to one of the 11 centers for assessment of FGFR-TACC expression by RNA analysis..

Patients will receive AZD4547 at a dose of 80mg bd on a continuous schedule, until disease progression. With the following hypothesis: P0: PFS6=15%, P1: PFS6=35%, with alpha=5% and power=80%, an initial cohort of 12 patients will be treated. If objective anti-tumor effects are observed, the cohort will be expanded to include a total number of 38 subjects. Grade II gliomas are also eligible but they will constitute an extra small cohort.

ELIGIBILITY:
Inclusion criteria:

1. Recurrent glioma after standard treatment, expressing the FGFR3-TACC3 or FGFR1-TACC1 fusion gene as confirmed by RT-PCR sequencing.
2. First recurrence occurring more than three months from the end of the radiotherapy or occurring outside the irradiated volume.
3. World Health Organisation performance status 0-2 (KPS>50) with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.
4. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.

   If a patient declines to participate in any voluntary exploratory research component of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study
5. Aged at least 18 years.
6. Patients should be using adequate contraceptive measures which should be maintained during the whole duration of AZD4547 treatment and at least 7 days after treatment suspension. Females should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation

Exclusion criteria:

1. Treatment with any of the following:

   * Nitrosourea within 6 weeks before the first dose of study treatment
   * Any investigational agents or study drugs from a previous clinical study within 30 days before the first dose of study treatment
   * Any other chemotherapy, anticancer immunotherapy or anticancer agents within 4 weeks before the first dose of study treatment, except hormonal therapy.
   * Potent inhibitors or inducers of CYP3A4 or 2D6 or substrates of CYP3A4 within the required washout period as specified in the section 7.3
   * Prior treatment in this or another AZD4547 study, or prior randomisation in a study in which AZD4547 is/was under investigation. Prior treatment with any FGFR inhibitor.
2. Major surgery (excluding placement of vascular access) within 14 days before the first dose of study treatment
3. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment
4. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required
5. Any of the following cardiac criteria:

   * Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's correction.Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
   * History of myocardial infarction, unstable angina, stroke or transient ischemic attack within the last 6 months
6. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophile count <1.5 x 109/L
   * Platelet count <100 x 109/L
   * Haemoglobin <90 g/L
   * Alanine aminotransferase >2.5 times the upper limit of normal (ULN)
   * Aspartate aminotransferase >2.5 times ULN Total bilirubin >1.5 times ULN
   * Creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
   * Corrected calcium >ULN
   * Phosphate >ULN
7. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD4547
8. History of hypersensitivity to active or inactive excipients of AZD4547 or drugs with a similar chemical structure or class to AZD4547
9. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
10. Any of the following ophthalmological criteria:

    * Current evidence or previous history of retinal pigmented epithelium detachment (RPED)
    * Previous laser treatment or intra-ocular injection for treatment of macular degeneration
    * Current evidence or previous history of dry or wet age-related macular degeneration
    * Current evidence or previous history of retinal vein occlusion (RVO)
    * Current evidence or previous history of retinal degenerative diseases (eg, hereditary)
    * Current evidence or previous history of any other clinically relevant chorioretinal defect
11. Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival measured according to RANO (Response Assessment in Neuro-Oncology) criteria | 6 months
  To assess the efficacy of AZD4547 by measuring the rate of Progression Free Survival at 6 months (PFS6) in recurrent malignant glioma patients with FGFR-TACC fusion.

SECONDARY OUTCOMES:
Overall response rate measured according to RANO criteria | 6 months
  To further assess the anti-tumor activity of AZD4547 for patients with recurrent glioma with FGFR-TACC fusion based on Overall Response Rate for patients with a measurable residue.
Duration of PFS | 12 months
  To further assess the anti-tumor activity of AZD4547 for patients with recurrent glioma with FGFR-TACC fusion based on the duration of PFS
Overall survival | 12 months
  To further assess the anti-tumor activity of AZD4547 for patients with recurrent glioma with a FGFR-TACC fusion based on Overall Survival AZD4547
Safety of AZD4547 (Number of patients who experienced grade III-IV (CTCAE v4.0) toxicity related to the drug) | 6 months
Pharmacokinetic of AZD4547: Maximum Plasma Concentration [Cmax] | Dosages will be performed at the cycle 2 or 3: predose, 2, 3, 4 and 6h post-dose
Pharmacokinetic of AZD4547: Area Under the Curve [AUC]). | Dosages will be performed at the cycle 2 or 3: predose, 2, 3, 4 and 6h post-dose
Pharmacokinetic of AZD4547: Residual Plasma Concentration | Dosages will be performed at the cycle 2 or 3: predose, 2, 3, 4 and 6h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sanson, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Neuro onsology unit - Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No